CLINICAL TRIAL: NCT03195699
Title: Phase I Study of TTI-101, an Oral Inhibitor of Signal Transducer and Activator of Transcription (STAT) 3, in Patients with Advanced Cancers
Brief Title: Oral STAT3 Inhibitor, TTI-101, in Patients with Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tvardi Therapeutics, Incorporated (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SM_CP2016-0842
Record Dates: First submitted 2017-06-09; First posted 2017-06-22 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Head and Neck Squamous Cell Carcinoma; Non Small Cell Lung Cancer; Hepatocellular Cancer; Colorectal Cancer; Gastric Adenocarcinoma; Melanoma; Advanced Cancer
Keywords: STAT3, cancer, inhibitor, advanced cancer
MeSH Terms: conditions — Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Liver Neoplasms; Colorectal Neoplasms; Melanoma; Neoplasms | interventions — C188-9 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose escalation study (Experimental): Participants will receive up to 4 dose levels of TTI-101 to determine RP2D
  Interventions: Drug: TTI-101
- Dose expansion study (Experimental): Enrollment in the dose expansion may commence with approval from the safety review committee. Participants will be enrolled and treated at the RP2D of TTI-101
  Interventions: Drug: TTI-101
- Food effect study (Experimental): Participants will be treated with TTI-101 at the RP2D under fed and fasted conditions to assess the bioavailability of TTI-101 and to determine the best conditions for taking the study drug
  Interventions: Drug: TTI-101
- Dose expansion, cross-over study (Experimental): Participants will be administered different formulations of TTI-101 to compare bioavailability.
  Interventions: Drug: TTI-101

INTERVENTIONS:
Drug: TTI-101 — Oral capsule
Drug: TTI-101 — Oral tablet
  Arms: Dose expansion, cross-over study

SUMMARY:
Many patients have cancers that have increased activity of a protein called STAT3 that contributes critically to the development and growth of their cancer. Despite our knowledge of STAT3's importance to cancer, scientists and doctors have not developed a drug that targets it and that patients can take to treat their cancer more effectively than treatments that are now available. Tvardi Therapeutics, Incorporated has developed a compound, TTI-101, which can be given by mouth and acts as a direct inhibitor of STAT3. Administration of TTI-101 to mice demonstrated that it blocked growth of cancers of the breast, head and neck, lung, and liver and it was safe when administered at high doses to mice, rats, and dogs. In this application, Tvardi is proposing to further develop TTI-101 for treatment of solid tumors for which the prognosis is dismal. The investigators will determine how safe it is when administered to patients with cancer, determine whether an adequate dose can be administered to patients with cancer that will block STAT3 in their cancer, and determine whether treatment with TTI-101 leads to reduced growth of their cancer.

DETAILED DESCRIPTION:
Signal transducer and activator of transcription 3 (STAT3) is a member of a family of seven closely related proteins responsible for transmission of peptide hormone signals from the extracellular surface of cells to the nucleus. STAT3 is a master regulator of most key hallmarks and enablers of cancer, including cell proliferation, resistance to apoptosis, metastasis, immune evasion, tumor angiogenesis, epithelial mesenchymal transition (EMT), response to DNA damage, and the Warburg effect. STAT3 also is a key mediator of oncogene addiction and supports the self-renewal of tumor-initiating cancer stem cells that contribute to cancer initiation, cancer maintenance, and relapse in several types of tumors. STAT3 activity is increased in ~50% of all cancers, due either to naturally occurring STAT3 mutations, as have been demonstrated in human inflammatory hepatocellular adenomas and large granular lymphocytic leukemia, or, more commonly as a result of activation of signaling molecules upstream of STAT3, including receptor tyrosine kinases (RTK; e.g. epidermal growth factor receptor, EGFR), tyrosine kinase-associated receptors (e.g. the family of IL-6 cytokine receptors or G-protein coupled receptors, GPCR), and Src kinases (e.g. Src, Lck, Hck, Lyn, Fyn, or Fgr). Thus, STAT3 is an attractive target for drug development to treat many types of cancer including breast cancer, head and neck squamous cell carcinoma (HNSCC), non-small cell lung cancer (NSCLC), hepatocellular carcinoma (HCC), colorectal cancer (CRC), gastric adenocarcinoma and melanoma.

ELIGIBILITY:
Inclusion Criteria

All of the following inclusion criteria must be fulfilled for eligibility:

1. Age ≥18 years;
2. For patients with solid tumors (not unresectable HCC): Patients with histologically confirmed diagnosis of locally-advanced, inoperable, metastatic and/or treatment refractory solid tumors for whom there are no available therapies that will confer clinical benefit;
3. For patients with unresectable HCC: Patients with histologically confirmed diagnosis of locally advanced, inoperable, unresectable HCC who have failed first and second lines of therapy and Child-Pugh is A or beyond second line if the performance status is preserved and Child-Pugh is A.
4. Eastern Cooperative Oncology Group Performance status 0-1;
5. Hemoglobin ≥9.0 g/dL, neutrophil count ≥1.0 x 109/l, platelets ≥75 x 109/L;
6. Adequate renal function capability, as calculated by creatinine clearance >40 ml/min using the Cockroft-Gault formula;
7. Adequate liver function defined as total bilirubin <1.5 x ULN, and aspartate aminotransferase (AST)/alanine aminotransferase (ALT) <3 x ULN. For subjects with liver involvement, AST/ALT <5 x ULN; For subjects with liver involvement, AST/ALT <5 x ULN;
8. Measurable disease using clinically appropriate criteria for the type of malignancy, RECIST v 1.1 for solid tumors;
9. Negative pregnancy test at the screening visit for women of childbearing potential, defined as: female subjects after puberty unless they have been postmenopausal for at least two years, are surgically sterile, or are sexually inactive and will remain so for the course of the trial;
10. Willingness to avoid pregnancy and breast feeding beginning two weeks before the first TTI-101 dose and ending three months after the last trial treatment. Male subjects with female partners of childbearing potential and female subjects of childbearing potential must use adequate contraception in the judgment of the Investigator, such as a two-barrier method or a one-barrier method with spermicide or intrauterine device during trial treatment dosing and for 3 months after the last dose of the study; and
11. Ability to read and understand the informed consent form and willingness and ability to give informed consent and demonstrate comprehension of the trial before undergoing any trial activities.

Exclusion Criteria

Subjects are ineligible to enroll in this trial if they fulfill any of the following exclusion criteria:

1. Previous therapy with:

   1. Standard therapy including chemotherapy, immunotherapy, biologic therapy, or any other anticancer therapy within 28 days (or five elimination half-lives for non-cytotoxic drugs, whichever is shorter) of Day 1 of trial drug treatment (6 weeks for nitrosureas or mitomycin);
   2. Any investigational agent within 28 days of Day 1 of trial drug treatment or 5 half-lives for a small molecule/targeted therapy;
2. Extensive prior radiotherapy on more than 30% of bone marrow reserves, or prior bone marrow/stem cell transplantation within 5 years from enrollment; Ongoing toxicity (except alopecia) due to a prior therapy, unless returned to baseline or Grade 1 or less;
3. Major surgical intervention or participation in a therapeutic clinical trial within 28 days from Day 1 of the first dose of TTI-101;
4. Significantly impaired cardiac function such as unstable angina pectoris, congestive heart failure with New York Heart Association (NYHA) class III or IV, myocardial infarction within the last 12 months prior to trial entry; signs of pericardial effusion, serious arrhythmia (including QTc prolongation of >470 ms and/or pacemaker) or prior diagnosis of congenital long QT syndrome or left ventricular ejection fraction <50% on screening echocardiogram;
5. History of cerebral vascular accident or stroke within the previous 2 years;
6. Uncontrolled hypertension (>160/100mm Hg);
7. History of Grade 3 or 4 allergic reactions attributed to compounds of similar chemical or biologic composition as TTI-101 (hydroxyl-naphthalene sulfonamides);
8. Known active metastases in the central nervous system (unless stable by brain imaging studies for at least 1 month without evidence of cerebral edema and no requirements for corticosteroids or anticonvulsants);
9. History of difficulty swallowing, malabsorption, or other chronic gastrointestinal disease or conditions that may hamper compliance and/or absorption of the investigational product;
10. Known human immunodeficiency virus (HIV);
11. Subjects with chronic hepatitis B virus (HBV) infection, unless screening viral load <100 IU/mL on stable doses of antiviral therapy. Note: Subjects with chronic HCV infection are allowed to enroll in the study but do not have a defined maximum viral load requirement for study entry;
12. Legal incapacity or limited legal capacity;
13. Pregnant or lactating women;
14. Any other condition, which in the opinion of the investigator, might impair the subject's tolerance of trial treatment, the safety of the individual subject, or the outcome of the trial;
15. Previous treatment of the current malignancy with a STAT inhibitor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of TTI-101 | 28 days
  To determine the maximum tolerated dose (MTD), dose-limiting toxicities, and tolerability of TTI-101 administered orally to patients with advanced breast cancer and other solid tumors. Dose-limiting toxicity is defined as a Grade 3 or above adverse event (using CTCAE v5.0) within the first treatment cycle (28-days).
Pharmacokinetics - Cmax | 18 months
  Cmax(obs) will be determined by direct inspection of the plasma drug concentration versus time data point values.
Pharmacokinetics - Tmax | 18 months
  Tmax(obs) will also be determined by direct inspection of the plasma drug concentration versus time data point values.
Pharmacokinetics - AUC(0-t) | 18 months
  AUC(0-t) (where t = the time point for the last sample on the pharmacokinetic profile in which quantifiable drug was detected) will be estimated using linear or linear/log trapezoidal calculation.

SECONDARY OUTCOMES:
Pharmacodynamics of TTI-101 in patients | 18 months
  Levels of pY-STAT3 measured before and before and after receiving TTI-101 will be measured.
Complete Response (CR) - Target Lesions | 18 months
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
Partial Response (PR) - Target Lesions | 18 months
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Progressive Disease (PD) - Target Lesions | 18 months
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Stable Disease (SD) - Target Lesions | 18 months
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Complete Response (CR) - Non-target Lesions | 18 months
  Complete Response (CR): Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
Non-CR/Non-PD - Non-target Lesions | 6 months
  Non-CR/Non-PD: Persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits.
Progressive Disease (PD) - Non-target Lesions | 18 months
  Progressive Disease (PD): Unequivocal progression of existing non-target lesions. (Note: the appearance of one or more new lesions is also considered progression).
Best Overall Response | 18 months
  The best overall response is the best response recorded from the start of the study treatment until the end of treatment, taking into account any requirement for confirmation. The patient's best overall response assignment will depend on the findings of both target and non-target disease and will also take into consideration the appearance of new lesions.

OTHER OUTCOMES:
Explore association between biomarkers and antitumor efficacy and survival outcome based on RECIST 1.1 for uHCC patients. | 18 months
  Assess the association between STAT3 inhibition, fibrosis (if applicable), antitumor activity and survival outcomes after receiving TTI-101. Tissue and blood immune monitoring will be based on 2 biopsies. Association between biomarkers including pY-STAT3, PD1, and PD-L1 proteins expression by IHC, gene expression profiling, and antitumor efficacy and survival outcome of TTI-101 based on RECIST 1.1.
Assess the effect of food on bioavailability | 18 months
  Assess the effect of food on bioavailability of TTI-101 in the dose expansion phase
Assess the bioavailability between different formulations of TTI-101 | 18 months
  Assess the bioavailability between different formulations of TTI-101 in the dose expansion phase

CONTACTS AND LOCATIONS:
Overall Officials: Apostolia Tsimberidou, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Mays Cancer Center at University of Texas Health Science Center SA, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsimberidou AM, Vining DJ, Arora SP, de Achaval S, Larson J, Kauh J, Cartwright C, Avritscher R, Alibhai I, Tweardy DJ, Kaseb AO. Phase I Trial of TTI-101, a First-in-Class Oral Inhibitor of STAT3, in Patients with Advanced Solid Tumors. Clin Cancer Res. 2025 Mar 17;31(6):965-974. doi: 10.1158/1078-0432.CCR-24-2920. PMID 39792482